CLINICAL TRIAL: NCT03514121
Title: A Phase 1a/1b Study of FPA150, an Anti-B7-H4 Antibody, in Patients With Advanced Solid Tumors
Brief Title: FPA150 in Patients With Advanced Solid Tumors
Acronym: FPA150-001
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The Sponsor terminated the study for reasons unrelated to safety.
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPA150-001
Record Dates: First submitted 2018-03-27; First posted 2018-05-02 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Ovarian Cancer; Endometrial Cancer; Advanced Solid Tumors
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single arm trial with multiple cohorts
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1a dose escalation/1b dose expansion (Experimental): The study consists of Phase 1a dose escalation, Phase 1a dose exploration, Phase 1a combination safety-lead-in and Phase 1b dose expansion
  Interventions: Biological: FPA150; Biological: Pembrolizumab

INTERVENTIONS:
Biological: FPA150 — A monoclonal antibody against B7-H4
Biological: Pembrolizumab — An anti-PD1 antibody

SUMMARY:
This is a multi-center study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy of FPA150, an anti-B7H4 antibody alone or in combination with pembrolizumab an anti-PD1 antibody in patients with advanced solid tumors. The Phase 1a, open-label, cohort will identify a recommended dose of FPA150 to use for Phase 1a Combination (FPA150 and Pembrolizumab) Safety Lead-in and for Phase 1b monotherapy cohorts.

DETAILED DESCRIPTION:
This is a Phase 1a/1b open-label, multicenter study to evaluate the dosing, safety, tolerability, PK, pharmacodynamics, and preliminary efficacy of FPA150 as monotherapy and in combination with pembrolizumab, an anti-PD1 antibody, in patients with advanced solid tumors.

This study includes a Phase 1a FPA150 Monotherapy Dose Escalation, Phase 1a Monotherapy Dose Exploration, Phase 1a combination Safety Lead-in (FPA150 + pembrolizumab), a Phase 1b FPA150 Monotherapy Dose Expansion, and a Phase 1b combination Dose Expansion (FPA150 + pembrolizumab).

The Phase 1a Monotherapy Dose Escalation will include an initial accelerated titration design followed by a standard 3+3 dose escalation design until the MTD and/or RD for Phase 1b is determined. The Phase 1a combination Safety Lead-In will start enrolling once the FPA150 monotherapy RD is identified in Phase 1a monotherapy dose escalation and will continue until the FPA150 MTD/RD in combination is identified. Phase 1a FPA150 monotherapy Dose Exploration may include cohorts that may enroll beyond 3 patients whose tumors express high levels of B7-H4 protein and/or have varying levels of B7H4 expression including low (<10% IHC 2+ or 3+ scores) or no expression on their tumor cells (up to 20 additional patients across all dose levels) to further evaluate safety, PK, pharmacodynamics, and clinical activity at that dose (to be conditional upon the dose level clearing DLT criteria).

Phase 1b will be the Dose Expansion (monotherapy and combination) portion of the study.

Enrollment into Phase 1b Dose Expansion will begin after identification of the MTD and/or RD in Phase 1a (monotherapy and Safety Lead-in). Preliminary efficacy will be evaluated in Phase 1b in planned expansion cohorts that include patients with specific tumor types that are B7-H4+ advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria (Phase 1a Monotherapy and Combination Therapy):

* Histologically confirmed solid tumors except primary central nervous system (CNS) tumors.
* Disease that is unresectable, locally advanced, or metastatic.
* Patients must have had progressive disease during or after, or refused, appropriate standard therapy for their tumor type.
* All patients must have at least one measurable lesion at baseline according to RECIST v1.1; tumor sites situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
* Adequate washout for prior anti-cancer therapy (ie, ≥ 5 half-lives or 4 weeks since the last dose, whichever is shorter).
* Availability of archival tumor tissue and consent to providing archival tumor for retrospective biomarker analysis, or willingness to undergo a fresh tumor biopsy during screening (a biopsy is required for patients in the Phase 1a Dose Exploration portion).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Prior radiotherapy must be completed at least 2 weeks before the first dose of study drug.
* Prior radiopharmaceuticals (eg strontium, samarium) must be completed at least 8 weeks before the first dose of study drug.
* Prior surgery requiring general anesthesia must be completed one week before first study drug administration. Surgery requiring local/epidural must be completed at least 72 hours before first study drug administration.
* Screening laboratory values must meet the following criteria:

  * Neutrophils ≥ 1200 cells/ µL
  * Platelets ≥ 75 × 103/ µL
  * Hemoglobin (Hb) ≥ 9.0 g/dL
  * Serum creatinine < 1.5× ULN or creatinine clearance (CrCl) of ≥ 40 mL/ minute
  * AST and ALT < 3× ULN (<5ULN in patients with liver metastases)
  * Bilirubin < 1.5× ULN (except patients with Gilbert's syndrome, who must have total bilirubin < 3 mg/dL)
* For Phase 1a Combination Safety Lead-in Patients ONLY:

  * B7-H4 positive ovarian cancer
  * or cytologically confirmed diagnosis of recurrent epithelial ovarian, primary peritoneal, or fallopian tube carcinoma that is refractory to existing therapy(ies) known to provide clinical benefit
  * Progressive disease on or after at least two prior regimens of treatment including at least one platinum-containing regimen, or unable to tolerate additional chemotherapy
  * No prior therapy with an anti-PD1 or PD-L1-directed agent

Inclusion Criteria (Phase 1b monotherapy and combination):

* All Inclusion Criteria for Phase 1a (Exception: Phase 1a Inclusion Criterion #1).
* Positive for B7-H4 expression in an archival or fresh tumor sample as evaluated by an accompanying validated central laboratory IHC assay. Archival tissue for patients enrolled in Cohort 1b1 (Breast Cancer) must be within 24 months prior to pre-screening.
* History of other malignancy is permitted provided it has been definitively treated with no evidence of recurrence within the past 2 years (Exception: Definitively treated non-melanoma skin cancer, lobular cancer in situ, and cervical cancer in situ within 2 years are permitted). Cohort Specific Phase 1b Criteria (monotherapy and combination therapy)

Breast Cancer Cohorts:

TNBC:

* Histologically or cytologically confirmed metastatic TNBC
* At least two prior lines of systemic chemotherapy with at least one being administered in the metastatic setting

HR+ Breast:

* Histologically or cytologically confirmed metastatic HR+ breast carcinoma
* Patients must have received at least two prior lines of hormonal therapy
* Patients must have received at least one prior line of systemic chemotherapy (in the adjuvant or metastatic setting)

Ovarian Cancer (monotherapy):

* Histologically or cytologically confirmed diagnosis of recurrent epithelial ovarian, primary peritoneal, or fallopian tube carcinoma that is refractory to existing
* Progressive disease on or after at least two prior regimens of treatment including at least one platinum-containing regimen, or unable to tolerate additional chemotherapy

Endometrial Cancer:

* Histologically or cytologically confirmed recurrent or persistent endometrial cancer that is refractory to curative or established treatments
* Progressive disease on or after at least one prior regimen of systemic chemotherapy, or unable to tolerate systemic chemotherapy

Ovarian Cancer (combination):

Histologically or cytologically confirmed diagnosis of recurrent epithelial ovarian, primary peritoneal, or fallopian tube carcinoma that is refractory to existing

* Progressive disease on or after at least two prior regimens of treatment including at least one platinum-containing regimen, or unable to tolerate additional chemotherapy
* No prior therapy with an anti-PD1 or PD-L1-directed agent

Exclusion Criteria:

* Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses > 10 mg/day prednisone or equivalent daily) must be discontinued at least 2 weeks before the first dose of study drug. Short courses of high dose steroids or continuous low dose (prednisone < 10 mg/day ) are allowed.
* Decreased cardiac function with New York Heart Association (NYHA) > Class 2 at screening.
* Uncontrolled or significant heart disorder such as unstable angina.
* QT interval corrected for heart rate (QTc) per institutional guidelines > 450 msec for males or > 470 msec for females at screening.
* Current unresolved infection or history of chronic, active, clinically significant infection (viral, bacterial, fungal, or other) which, in the opinion of the Investigator, would preclude the patient from exposure to a biologic agent or may pose a risk to patient safety.
* Any uncontrolled medical condition or psychiatric disorder which, in the opinion of the Investigator, would pose a risk to patient safety or interfere with study participation or interpretation of individual patient results.
* Active, known, or suspected autoimmune disease. Patients with Type I diabetes mellitus, hypothyroidism requiring only hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger, are permitted to enroll.
* Known history of testing positive for human immunodeficiency virus (HIV) 1 or 2 or known acquired immunodeficiency syndrome (AIDS).
* Positive test for hepatitis B virus surface antigen (HBsAg) or detectable hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection.
* Ongoing adverse effects from prior treatment > Grade 1 (with the exception of Grade 2 alopecia or peripheral neuropathy) based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
* Symptomatic interstitial lung disease or inflammatory pneumonitis.
* Untreated or active CNS or leptomeningeal metastases. Patients are eligible if metastases have been treated and patients are neurologically returned to baseline or neurologically stable (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks before the first dose of study drug.
* Evidence of coagulopathy or bleeding diathesis. Patients receiving stable therapeutic doses of anti-coagulants will be permitted.
* Transfusion of blood or platelets completed within 72 hours before the first dose of study drug.
* Any uncontrolled inflammatory GI disease including Crohn's Disease and ulcerative colitis
* For Cohort 1b1 only: Patients with HER2 positive disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (18):
- United States (13):
  - Honor Health, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Medical Oncology Associates, PS, Spokane, Washington
- South Korea (5):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Severance Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Samsung Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 25 study centers in the United Studies and the Republic of Korea, and participated from 27 March 2018 to 21 April 2021.
Groups:
- Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A: Participants with advanced solid tumors received FPA150 once every 3 weeks (Q3W) in escalating doses (Dose A-H) until the maximum tolerated dose (MTD) and/or recommended dose (RD) for Phase 1b was determined.
- Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B; Phase 1a Monotherapy Dose Escalation + Exploration Dose C; Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D; Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E; Phase 1a Monotherapy Dose Escalation + Exploration Dose F; Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G; Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H: Participants with advanced solid tumors received FPA150 Q3W in escalating doses until MTD and/or RD for Phase 1b was determined.
- Phase 1b Monotherapy FPA150 Dose H: Participants with breast, ovarian, or endometrial cancer received FPA150 MTD/RD.
- Phase 1a Combination Safety Lead-In & Phase 1b Combination FPA150 Dose H & Pembrolizumab 200 mg: Participants with ovarian cancer received FPA 150 Dose H in combination with pembrolizumab 200 mg IV Q3W during the Phase 1a Safety Lead-in. Participants with ovarian cancer in the Phase 1b Combination received FPA 150 Dose H in combination with pembrolizumab 200 mg IV Q3W.
Period: Overall Study
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H | Phase 1b Monotherapy FPA150 Dose H | Phase 1a Combination Safety Lead-In & Phase 1b Combination FPA150 Dose H & Pembrolizumab 200 mg
Started | 1 | 1 | 3 | 1 | 3 | 8 | 8 | 4 | 54 (Participants in 1b Monotherapy were stratified by cancer type for some data analysis, but they were not considered separate randomization groups.) | 12
Received Any Study Treatment | 1 | 1 | 3 | 1 | 3 | 8 | 8 | 4 | 54 | 12
1b Monotherapy (Breast) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0
1b Monotherapy (Ovarian) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
1b Monotherapy (Endometrial) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0
Phase 1a Combination Safety Lead-In | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Phase 1b Combination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Completed | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Not Completed | 0 | 1 | 2 | 0 | 2 | 7 | 7 | 4 | 53 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 7 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 26 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 1 | 2 | 3 | 2 | 7 | 3
Not completed — Study termination by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 3
Not completed — Investigator decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data from the safety population dataset (SAS) which included all participants who received any portion of at least one dose of FPA150.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H | Phase 1b Monotherapy FPA150 Dose H | Phase 1a Combination Safety Lead-In & Phase 1b Combination FPA150 Dose H & Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 8 | 8 | 4 | 54 | 12 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 1 | 1 | 4 | 4 | 3 | 33 | 6 | 54
  >=65 years | 0 | 1 | 2 | 0 | 2 | 4 | 4 | 1 | 21 | 6 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 2 | 5 | 7 | 3 | 54 | 12 | 88
  Male | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 6
  Not Hispanic or Latino | 1 | 0 | 2 | 1 | 3 | 7 | 7 | 3 | 53 | 12 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 13 | 1 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 5
  White | 0 | 1 | 3 | 1 | 3 | 8 | 6 | 2 | 38 | 10 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a Monotherapy: Number of Participants Experiencing Grade 3 and Grade 4 Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation subject that was administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment. Grade 3 and 4 severity ratings were defined as follows:
  Grade 3: Severe or medically significant but non-immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; severe AE Grade 4: Life-threatening consequences; urgent intervention indicated
Time Frame: From day 1 up to 28 days after last dose (median [min, max] treatment duration= 9.143 [3.00, 52.00] weeks)
Population: SAS: All participants who have received any portion of at least one dose of FPA150.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 8 | 8 | 4
Participants | 1 | 1 | 3 | 1 | 1 | 4 | 5 | 1

2. Primary Outcome: Phase 1a Monotherapy: Number of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as any of the following events regardless of attribution (except for those events clearly due to the underlying disease or extraneous causes):
  Any Grade 3 or higher non-hematologic toxicity (except Grade 3 nausea, vomiting, and diarrhea) that occurred within the first 21 days of treatment.
  Grade 3 nausea, vomiting, diarrhea lasting >72 hours, that occurred within the first 21 days of treatment.
  Febrile neutropenia and/or documented infection, Grade 4 neutropenia that lasted more than 7 days, Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia accompanied by bleeding within first 21 days of treatment.
  Aspartate aminotransferase (AST) / alanine transaminase (ALT) >3 × upper limit of normal (ULN) and concurrent total bilirubin > 2 × ULN that was not related to liver involvement with cancer.
  Other Grade 3 laboratory values that did not resolve within 72 hours. Any Grade 4 laboratory value regardless of clinical sequelae
Time Frame: Up to 21 days
Population: SAS: All participants who have received any portion of at least one dose of FPA150.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 8 | 8 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 1a Monotherapy: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as an AE that began or worsened in severity after at least one dose of study treatment (FPA150) had been administered. Clinically significant laboratory abnormalities and ECG abnormalities are included as TEAEs.
Time Frame: From day 1 up to 28 days after last dose (median [min, max] treatment duration= 9.143 [3.00, 52.00] weeks)
Population: SAS: All participants who have received any portion of at least one dose of FPA150.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 8 | 8 | 4
Participants | 1 | 1 | 3 | 1 | 3 | 7 | 7 | 4

4. Primary Outcome: Phase 1b Monotherapy: Number of Participants Experiencing AEs
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation subject that was administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment. A serious AE is defined as any AE that resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality/birth defect or important medical events. Clinically significant laboratory abnormalities and ECG abnormalities were included as TEAEs.
Time Frame: From day 1 up to 28 days after last dose (median [min, max] treatment duration= 6.35 [3.00, 108.14] weeks)
Population: SAS: All participants who have received any portion of at least one dose of FPA150.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Monotherapy: Participants with breast, ovarian, or endometrial cancer received FPA150 20mg/kg Q3W.
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 54
Participants
  Breast Cancer: number analyzed (Participants) | 21
  Breast Cancer | 18
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 16
  Endometrial Cancer: number analyzed (Participants) | 16
  Endometrial Cancer | 16

5. Primary Outcome: Phase 1a Combination Safety Lead-In & Phase 1b Combination: Number of Participants Experiencing AEs
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation subject that was administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment. A serious AE is defined as any AE that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect or important medical events that do not meet the preceding criteria but based on appropriate medical judgment may jeopardize the participant or may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: From day 1 up to 28 days after last dose (median [min, max] treatment duration= 12.00 [6.00, 36.43] weeks)
Population: SAS: All participants who have received any portion of at least one dose of FPA150.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1a Combination Safety Lead-In & Phase 1b Combination: Participants in Phase 1a received a combination of FPA150 20mg/kg and pembrolizumab 200mg Q3W. If DLTs were observed the dose of FPA150 was reduced.
  Participants in Phase 1b received FPA150 20mg/kg in combination with pembrolizumab 200mg Q3W.
Arm/Group | Phase 1a Combination Safety Lead-In & Phase 1b Combination
Number analyzed (Participants) | 12
Participants | 11

6. Primary Outcome: Phase 1a Combination Safety Lead-In & Phase 1b Combination: Number of Participants Experiencing Grade 3 and Grade 4 AEs
Description: as for outcome 5
Time Frame: From day 1 up to 28 days after last dose (median [min, max] treatment duration= 12.00 [6.00, 36.43] weeks)
Population: SAS: All participants who have received any portion of at least one dose of FPA150.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1a Combination Safety Lead-In & Phase 1b Combination: Participants in Phase 1a received a combination of FPA150 20mg/kg and pembrolizumab 200mg Q3W. If DLTs were observed the dose of FPA150 was reduced.
  Participants in Phase 1b received a combination of FPA150 20mg/kg in combination with pembrolizumab 200mg Q3W.
Arm/Group | Phase 1a Combination Safety Lead-In & Phase 1b Combination
Number analyzed (Participants) | 12
Participants | 4

7. Secondary Outcome: Phase 1a Monotherapy: Number of Participants With ADAs to FPA150
Description: All ADA samples were collected prior to dosing. A baseline ADA-positive patient was defined as a patient who had an ADA positive sample at baseline. Postbaseline treatment induced ADA positive is derived as participants with ADA negative at baseline and ADA positive at any postbaseline timepoint, or ADA positive at baseline and ADA positive with titer of at least 4-fold of the baseline titer at one or more postbaseline timepoint.
Time Frame: From day 1 up to 28 days after last dose (median [min, max] treatment duration= 9.143 [3.00, 52.00] weeks)
Population: ADA Analysis Set: The ADA Analysis Set included all enrolled participants who received at least 1 dose of FPA150 and had at least 1 ADA sample drawn at any timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 3 | 5 | 4
Participants
  Baseline: ADA Positive | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Baseline: ADA Negative | 1 | 1 | 2 | 1 | 3 | 3 | 4 | 4
  Baseline: Not Evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Postbaseline: ADA Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Postbaseline: ADA Negative | 1 | 1 | 3 | 1 | 2 | 3 | 4 | 3
  Postbaseline: Not Evaluable | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

8. Secondary Outcome: Phase 1b Monotherapy: Number of Participants With ADAs to FPA150 at Baseline
Description: as for outcome 7
Time Frame: Cycle 1 day 1 pre-dose (baseline)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 54
Participants
  Breast Cancer: number analyzed (Participants) | 21
  Breast Cancer | 1
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 1
  Endometrial Cancer: number analyzed (Participants) | 16
  Endometrial Cancer | 1

9. Secondary Outcome: Phase 1b Monotherapy: Number of Participants With ADAs to FPA150 Postbaseline
Description: as for outcome 7
Time Frame: From day 1 up to 28 days after last dose (median [min, max] treatment duration= 6.35 [3.00, 108.14] weeks)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 54
Participants
  Breast Cancer: number analyzed (Participants) | 21
  Breast Cancer | 0
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 1
  Endometrial Cancer: number analyzed (Participants) | 16
  Endometrial Cancer | 1

10. Secondary Outcome: Phase 1b Monotherapy: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as the percentage of participants who achieved best overall response (BOR) of either complete response (CR) or partial response (PR) based on investigator assessment of tumor lesions per RECIST v1.1. The BOR was the best response documented from first dose until the end of study, first disease progression, death, or start of new anti-cancer therapy, whichever was earlier.
Time Frame: Up to approximately 24 months
Population: Efficacy-Evaluable Analysis Set: included all participants that received at least 1 dose of FPA150, had at least 1 postbaseline evaluable tumor assessment unless death or clinical progressive disease occurred prior to the first post baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 54
Participants
  Breast Cancer: number analyzed (Participants) | 21
  Breast Cancer | 0
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 1
  Endometrial Cancer: number analyzed (Participants) | 16
  Endometrial Cancer | 0

11. Secondary Outcome: Phase 1b Monotherapy: Duration of Response (DOR) Per RECIST v1.1
Description: DOR is defined as the time from first onset of response (CR or PR determined by the investigator per RECIST v1.1) that is subsequently confirmed until the onset of progressive disease or death from any cause, whichever comes first. Patients who were alive and progression-free at the time of data analysis were censored at the time of their last assessment for tumor response. DOR was estimated using the Kaplan-Meier method.
Time Frame: Up to approximately 24 months
Population: Efficacy-Evaluable Analysis Set: included all participants that received at least 1 dose of FPA150, had at least 1 postbaseline evaluable tumor assessment unless death or clinical progressive disease occurred prior to the first post baseline disease assessment. Only responders have been included in the analysis.
Measure: Number (90% Confidence Interval); unit: months
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 1
months | NA [NA to NA] — Given single responder these data not reported due to patient privacy concerns.

12. Secondary Outcome: Phase 1b Monotherapy: Progression-free Survival (PFS) Per RECIST v1.1
Description: PFS defined as time from the first dose of study treatment until the first documentation by the investigator of disease progression per RECIST v1.1 or death from any cause, whichever comes first. Patients who were alive and progression-free at the time of data analysis were censored at the time of their last assessment for tumor response.
Time Frame: Up to approximately 24 months
Population: as for outcome 10
Measure: Mean (90% Confidence Interval); unit: months
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 10
months | 1.40 [0.79 to 5.42]

13. Secondary Outcome: Phase 1b Combination: PFS Per RECIST v1.1
Description: as for outcome 12
Time Frame: Up to approximately 24 months
Population: No PFS data for Phase 1b combination was collected due to study early termination. Data for phase 1a were considered exploratory.
Groups:
- Phase 1b Combination: Participants in Phase 1b received FPA150 20mg/kg in combination with pembrolizumab 200mg Q3W.
Arm/Group | Phase 1b Combination
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 1b Combination: ORR Per RECIST v1.1
Description: as for outcome 10
Time Frame: Up to approximately 24 months
Population: No ORR data for Phase 1b combination was collected due to study early termination. Data for phase 1a were considered exploratory.
Arm/Group | Phase 1b Combination
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 1b Combination: DOR Per RECIST v1.1
Description: as for outcome 11
Time Frame: Up to approximately 24 months
Population: No DOR data for Phase 1b combination was collected due to study early termination. Data for phase 1a were considered exploratory.
Arm/Group | Phase 1b Combination
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase 1a Monotherapy: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of FPA150
Description: FPA150 concentration in serum was determined using an enzyme linked immunosorbent assay (ELISA) method and the PK parameters were derived from serum FPA150 concentration-time data using non-compartment analysis.
Time Frame: Cycle 1 (cycle = 21 days) day 1 pre-dose, 15min and 4h post-dose, day 2 (24h), day 4 (72h), day 8 (168h) post-dose, and day 15. Cycle 2, 3, 4 ,5 ,7, 9, day 1 pre-dose, day 1 (15min) post-dose. After cycle 9, day 1 every 4th dose (12 weeks) up to 52 weeks
Population: PK Analysis Population: All participants who received at least one dose of FPA150 and had at least one FPA150 serum concentration result. Only participants with available data are included. Participants with available data are included.
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 3 | 5 | 4
day*µg/mL | 0.7591 (NA) — Standard deviation not calculable from 1 participant analyzed. | 9.2670 (NA) — Standard deviation not calculable from 1 participant analyzed. | 8.2148 (0.21781) | 37.4379 (NA) — Standard deviation not calculable from 1 participant analyzed. | 136.6567 (38.99659) | 407.1698 (69.78823) | 1376.0347 (411.93171) | 2468.4741 (638.37831)

17. Secondary Outcome: Phase 1a Monotherapy: Time to Reach Maximum Serum Concentration (Tmax) of FPA150
Time Frame: as for outcome 16
Population: PK Analysis Population: All participants who received at least one dose of FPA150 and had at least one FPA150 serum concentration result. Only participants with available data are included.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 3 | 5 | 4
Days | 0.0521 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.2146 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.0549 (0.00184) | 0.0556 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.0998 (0.09405) | 0.0523 (0.01107) | 0.1449 (0.08381) | 0.0892 (0.07284)

18. Secondary Outcome: Phase 1a Monotherapy: Maximum Serum Concentration (Cmax) of FPA150
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 3 | 5 | 4
μg/mL | 0.0521 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.2146 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.0549 (0.00184) | 0.0556 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.0998 (0.09405) | 0.0523 (0.01107) | 0.1449 (0.08381) | 0.0892 (0.07284)

19. Secondary Outcome: Phase 1a Monotherapy: Trough Serum Concentration (Ctrough) of FPA150
Time Frame: as for outcome 16
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 3 | 5 | 4
µg/mL | 0.0000 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.1160 (NA) — Standard deviation not calculable from 1 participant analyzed. | 0.0000 (0.00000) | 0.6050 (NA) — Standard deviation not calculable from 1 participant analyzed. | 3.0825 (2.18567) | 9.5243 (5.17826) | 30.5385 (7.13748) | 37.9028 (4.28708)

20. Secondary Outcome: Phase 1a Monotherapy: Terminal Half-Life (T1/2) of FPA150
Time Frame: as for outcome 16
Population: Cycle 1 (cycle = 21 days) day 1 pre-dose, 15min and 4h post-dose, day 2 (24h), day 4 (72h), day 8 (168h) post-dose, and day 15. Cycle 2, 3, 4 ,5 ,7, 9, day 1 pre-dose, day 1 (15min) post-dose. After cycle 9, day 1 every 4th dose (12 weeks) up to 52 weeks
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 3 | 3 | 5 | 4
day | 2.7207 (NA) — Standard deviation not calculable from 1 participant analyzed. | 7.2128 (NA) — Standard deviation not calculable from 1 participant analyzed. | 4.6081 (0.99726) | 8.3932 (NA) — Standard deviation not calculable from 1 participant analyzed. | 10.4675 (3.25703) | 13.0391 (4.74220) | 8.3539 (2.80118) | 9.1097 (1.25064)

21. Secondary Outcome: Phase 1b Monotherapy: AUClast of FPA150
Time Frame: Cycle 1 (one cycle = 21 days) day 1 pre-dose, day 1 15min and 4h post-dose, day 2 (24h), day 4 (72h), day 8 (168h) post-dose, and day 15. Cycle 2, 3, 4 ,5 ,7, 9, day 1 pre-dose, day 1 (15min) post-dose. After cycle 9, day 1 every 4th dose (12 weeks)
Population: PK Analysis Population: All participants who received at least one dose of FPA150 and had at least one FPA150 serum concentration result.
Measure: Mean (Standard Deviation); unit: Day*µg/mL
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 54
Day*µg/mL
  Breast Cancer: number analyzed (Participants) | 21
  Breast Cancer | 2415.8123 (951.56795)
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 2664.4820 (761.19550)
  Endometrial Cancer: number analyzed (Participants) | 16
  Endometrial Cancer | 2785.3974 (941.95867)

22. Secondary Outcome: Phase 1b Monotherapy: Time to Reach Cmax of FPA150
Time Frame: Cycle 1 (cycle = 21 days) day 1 pre-dose, 15min and 4h post-dose, day 2 (24h), day 4 (72h), day 8 (168h) post-dose, and day 15. Cycle 2, 3, 4 ,5 ,7, 9, day 1 pre-dose, day 1 (15min) post-dose. After cycle 9, day 1 every 4th dose (12 weeks) up to 108 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 54
day
  Breast Cancer: number analyzed (Participants) | 21
  Breast Cancer | 0.0944 (0.06325)
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 0.1056 (0.06988)
  Endometrial Cancer: number analyzed (Participants) | 16
  Endometrial Cancer | 1.2803 (4.71147)

23. Secondary Outcome: Phase 1b Monotherapy: Cmax of FPA150
Time Frame: as for outcome 22
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 54
µg/mL
  Breast Cancer: number analyzed (Participants) | 21
  Breast Cancer | 383.8841 (89.76028)
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 422.5332 (101.20218)
  Endometrial Cancer: number analyzed (Participants) | 16
  Endometrial Cancer | 456.9944 (101.87663)

24. Secondary Outcome: Phase 1b Monotherapy: Cthrough of FPA150
Time Frame: as for outcome 22
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 49
µg/mL
  Breast Cancer: number analyzed (Participants) | 19
  Breast Cancer | 57.6900 (37.24538)
  Ovarian Cancer: number analyzed (Participants) | 16
  Ovarian Cancer | 56.1074 (27.88026)
  Endometrial Cancer: number analyzed (Participants) | 14
  Endometrial Cancer | 72.1686 (78.21933)

25. Secondary Outcome: Phase 1b Monotherapy: T1/2 of FPA150 in Days
Time Frame: as for outcome 22
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Phase 1b Monotherapy
Number analyzed (Participants) | 49
day
  Breast Cancer: number analyzed (Participants) | 17
  Breast Cancer | 9.3232 (2.63376)
  Ovarian Cancer: number analyzed (Participants) | 17
  Ovarian Cancer | 10.0294 (3.90951)
  Endometrial Cancer: number analyzed (Participants) | 15
  Endometrial Cancer | 7.9802 (3.72524)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 28 days after last dose of study drug. Median (min, max) duration of exposure was 9.14 [3.0, 52.0] weeks for the Phase 1a Dose Escalation + Explorations part of the study, 6.36 [3.0, 108.1] weeks for the Phase 1b Monotherapy part and 12.00 [6.0, 36.4] weeks for the Phase 1a combination lead-in and Phase 1b combination.
Groups:
- Phase 1b Monotherapy FPA150 Dose H (Breast); Phase 1b Monotherapy FPA150 Dose H (Ovarian); Phase 1b Monotherapy FPA150 Dose H (Endometrial): Participants with breast, ovarian, or endometrial cancer received FPA150 MTD/RD.
Arm/Group | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B | Phase 1a Monotherapy Dose Escalation + Exploration Dose C | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E | Phase 1a Monotherapy Dose Escalation + Exploration Dose F | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H | Phase 1b Monotherapy FPA150 Dose H (Breast) | Phase 1b Monotherapy FPA150 Dose H (Ovarian) | Phase 1b Monotherapy FPA150 Dose H (Endometrial) | Phase 1a Combination Safety Lead-In & Phase 1b Combination FPA150 Dose H & Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 0/1 | 0/3 | 3/8 | 2/8 | 1/4 | 9/21 | 10/17 | 7/16 | 3/12
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/3 | 0/1 | 1/3 | 1/8 | 3/8 | 0/4 | 3/21 | 6/17 | 5/16 | 3/12
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 1/1 | 3/3 | 7/8 | 7/8 | 4/4 | 16/21 | 14/17 | 16/16 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A (N=1) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B (N=1) | Phase 1a Monotherapy Dose Escalation + Exploration Dose C (N=3) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D (N=1) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E (N=3) | Phase 1a Monotherapy Dose Escalation + Exploration Dose F (N=8) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G (N=8) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H (N=4) | Phase 1b Monotherapy FPA150 Dose H (Breast) (N=21) | Phase 1b Monotherapy FPA150 Dose H (Ovarian) (N=17) | Phase 1b Monotherapy FPA150 Dose H (Endometrial) (N=16) | Phase 1a Combination Safety Lead-In & Phase 1b Combination FPA150 Dose H & Pembrolizumab 200 mg (N=12)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose A (N=1) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose B (N=1) | Phase 1a Monotherapy Dose Escalation + Exploration Dose C (N=3) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose D (N=1) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose E (N=3) | Phase 1a Monotherapy Dose Escalation + Exploration Dose F (N=8) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose G (N=8) | Phase 1a Monotherapy Dose Escalation + Exploration FPA150 Dose H (N=4) | Phase 1b Monotherapy FPA150 Dose H (Breast) (N=21) | Phase 1b Monotherapy FPA150 Dose H (Ovarian) (N=17) | Phase 1b Monotherapy FPA150 Dose H (Endometrial) (N=16) | Phase 1a Combination Safety Lead-In & Phase 1b Combination FPA150 Dose H & Pembrolizumab 200 mg (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 3 | 4 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye haematoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 4 | 3 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 4 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 2 | 4 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 1 | 1 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT03514121/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03514121/SAP_001.pdf